CLINICAL TRIAL: NCT00852566
Title: An Open-Label, Randomized, Multicenter Phase II Trial Comparing the Depletion of Malignant Stem Cells With Dasatinib vs. Imatinib in Patients With Newly Diagnosed Chronic Phase Chronic Myeloid
Brief Title: Randomized Study Comparing the Effect of Dasatinib and Imatinib on Malignant Stem Cells in Chronic Myeloid Leukemia
Acronym: NordCML006
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-004106-13
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; tyrosine kinase inhibitor; stem cell; Philadelphia chromosome; dasatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome | interventions — Imatinib Mesylate; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imatinib (Active Comparator): Standard treatment Imatinib 400mg OD
  Interventions: Drug: Imatinib
- dasatinib (Experimental): Dasatinib 100mg OD
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Imatinib — Per oral imatinib 400mg once daily (continuous medication)
  Other Names: Glivec
  Arms: Imatinib
Drug: Dasatinib — Per oral dasatinib 100mg once daily (continuous medication)
  Other Names: Sprycel
  Arms: dasatinib

SUMMARY:
A randomized multi-center study comparing the effect of dasatinib and imatinib on malignant stem cells in newly diagnosed chronic phase chronic myeloid leukemia (CML) patients. The research hypothesis is that treatment with dasatinib 100 mg daily (QD) results in greater and more rapid depletion of the Philadelphia (Ph) -positive stem cell pool within 6 months of therapy than imatinib 400 mg QD in newly diagnosed CML patients. The study duration is 18 months and approximately 40 patients will be recruited to the study.

DETAILED DESCRIPTION:
An Open-Label, Randomized, Multicenter Phase II Trial Comparing the depletion of malignant stem cells with Dasatinib vs. Imatinib in Patients with Newly Diagnosed Chronic Phase Chronic Myeloid Leukemia

Estimated Number of Study Centers and Countries/Regions: Appr. 12 sites in 5 Nordic countries. Stem cell analyses will be performed in 4 Nordic centers (Helsinki, Lund, Oslo and Stockholm).

Study Phase: II

Research Hypothesis: Treatment with dasatinib 100 mg daily (QD) results in greater and more rapid depletion of the Philadelphia (Ph) -positive stem cell pool within 6 months of therapy than imatinib 400 mg QD in newly diagnosed chronic phase (CP) chronic myeloid leukemia (CML) patients.

Primary Objective: To compare the number of Ph-positive cells in the stem cell compartment in newly diagnosed CP CML patients treated with dasatinib 100 mg QD vs. imatinib 400 mg QD.

Study Design: open-label randomized Phase II trial in newly diagnosed CML patients in CP. Patients will be randomized to receive dasatinib at a starting dose of 100 mg QD or imatinib at a starting dose of 400 mg QD.

Duration of Study: The study will be open for enrollment until the planned number of 40 patients is randomized. All patients will be treated and/or followed for up to 18 months. Based on the amendment 1 (Oct 2011), the follow-up of the patients will continue additional 4 years until 31.12.2015.

Number of Patients per Group: Approximately 40 patients will be randomized, 20 patients to dasatinib and 20 to imatinib. Additional patients will be recruited in case insufficient amount of representative samples have been obtained from first 40 patients.

Study Population: Patients 18 years or older with a newly diagnosed CP CML, not previously treated with any systemic treatments for CML

Study Assessments and Endpoints:

All stem cell assays are based on the preselection of CD34+ cells from large volume of bone marrow (BM) aspirates using paramagnetic beads. The CD34+ fraction will be further subdivided based on the expression of CD38 marker (positive vs. negative) using a sorting flow cytometer.

The primary endpoint is a comparison of proportion of Ph-positive cells in stem cell compartments (CD34+CD38neg and CD34+CD38+) at 6 months between the study arms.

Secondary endpoints are comparisons between treatment arms for: (1) the number of Ph-positive cells in all stem cell compartments at 1 and 3 months, (2) BCR-ABL RQ-PCR in blood at 1, 3, 6, 12 and 18 months, and (3) rate of CCyR within 3, 6, 12 and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients are able to provide written informed consent
* Patients must have CML in CP which is defined by the presence of all of the following criteria:

  * < 15% blasts in peripheral blood (PB) and BM.
  * < 30% blasts plus promyelocytes in PB and BM.
  * < 20% basophils in the PB.
  * ≥ 100 x 109/L platelets.
  * No evidence of extramedullary leukemia apart from hepatosplenomegaly
  * Ph+ or variants must be demonstrated by BM cytogenetics, FISH or PCR.
  * Previously untreated CML in CP, with the exception of hydroxyurea or anagrelide
* Patients must be enrolled in this study within 90 days after the date of first being diagnosed with CML
* ECOG Performance Status (PS) Score 0 - 1 (see Appendix 2)
* Adequate hepatic function defined as: total bilirubin ≤ 2.0 times the institutional upper limit of normal (ULN) in absence of Gilbert type unconjugated hyperbilirubinemia; alanine aminotransferase (ALAT≤ 2.5 times the institutional ULN.
* Adequate renal function defined as serum creatinine ≤ 2 times the institutional ULN.
* Men and women, ages 18 years and older.
* Adequate BM aspiration sample before the start of study treatment (i.e sample is sufficient for stem cell analysis)
* Potentially fertile women must use an adequate method of contraception to avoid pregnancy throughout the study.
* Potentially fertile women must have a negative serum or urine pregnancy test

Exclusion Criteria:

* Fertile women who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study
* Women who are pregnant or breastfeeding.
* Men with fertile sexual partners who can or will not use an acceptable contraception method for the entire study
* A serious uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy.
* Known pleural effusion at baseline.
* Uncontrolled or significant cardiovascular disease
* History of significant bleeding disorder unrelated to CML, including:
* Prior chemotherapy for peripheral stem cell mobilization.
* Inadequate BM aspiration sample due to marrow fibrosis or other reasons
* Prior or concurrent malignancy
* Severe psychiatric illness, imprisonment or mental impairment inflicting on ability to give informed consent
* Abuse of alcohol, prescribed or illicit drugs
* Evidence of digestive dysfunction that would prevent administration of study therapy by mouth.
* Prohibited Treatments and/or Therapies

  * Any prior treatment with interferon
  * Any prior treatment with dasatinib
  * Any prior treatment with imatinib
  * Any other prior systemic treatments, with anti-CML activity [except for anagrelide, or hydroxyurea (HU)].
* Patients currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes as described in Appendix 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Ph-positive cells in stem cell compartments | 6 months
  proportion of Ph-positive cells in stem cell compartments (CD34+CD38neg and CD34+CD38+)

SECONDARY OUTCOMES:
BCR-ABL RQ-PCR in blood | up to 18 months (1, 3, 6, 12 and 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Satu Mustjoki, MD, PhD, Principal Investigator — Helsinki University Central Hospital, helsinki, Finland; Henrik Hjorth-Hansen, MD, PhD, Study Chair — St. Olavs Hospital, Trondheim, Norway; Ole Weiss-Bjerrum, MD, PhD, Study Chair — Rigshospitalet, Denmark; Ingunn Dybedal, MD, PhD, Study Chair — Rikshospitalet, Oslo, Norway; Tobias Gedde-Dahl, MD, PhD, Study Chair — Rikshospitalet, Oslo, Norway; Kimmo Porkka, MD, PhD, Study Chair — Helsinki University Central Hospital, Helsinki, Finland; Johan Richter, MD, PhD, Study Chair — University of Lund, Lund, Sweden; Bengt Simonsson, MD, PhD, Study Chair — University Hospital, Uppsala, Sweden; Leif Stenke, MD, PhD, Study Chair — Karolinska Institutet
Locations (7):
- Helsinki University Central Hospital, Helsinki, Finland
- Norway (3):
  - Bergen University Central Hospital, Bergen
  - Rikshospitalet, Oslo
  - St. Olavs Hospital, Trondheim
- Sweden (3):
  - Lund University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

REFERENCES:
- [Result] Hjorth-Hansen H, Stenke L, Soderlund S, Dreimane A, Ehrencrona H, Gedde-Dahl T, Gjertsen BT, Hoglund M, Koskenvesa P, Lotfi K, Majeed W, Markevarn B, Ohm L, Olsson-Stromberg U, Remes K, Suominen M, Simonsson B, Porkka K, Mustjoki S, Richter J; Nordic CML Study Group. Dasatinib induces fast and deep responses in newly diagnosed chronic myeloid leukaemia patients in chronic phase: clinical results from a randomised phase-2 study (NordCML006). Eur J Haematol. 2015 Mar;94(3):243-50. doi: 10.1111/ejh.12423. Epub 2014 Sep 13. PMID 25082346
- [Derived] Christiansson L, Soderlund S, Mangsbo S, Hjorth-Hansen H, Hoglund M, Markevarn B, Richter J, Stenke L, Mustjoki S, Loskog A, Olsson-Stromberg U. The tyrosine kinase inhibitors imatinib and dasatinib reduce myeloid suppressor cells and release effector lymphocyte responses. Mol Cancer Ther. 2015 May;14(5):1181-91. doi: 10.1158/1535-7163.MCT-14-0849. Epub 2015 Mar 11. PMID 25761894
- [Derived] Mustjoki S, Richter J, Barbany G, Ehrencrona H, Fioretos T, Gedde-Dahl T, Gjertsen BT, Hovland R, Hernesniemi S, Josefsen D, Koskenvesa P, Dybedal I, Markevarn B, Olofsson T, Olsson-Stromberg U, Rapakko K, Thunberg S, Stenke L, Simonsson B, Porkka K, Hjorth-Hansen H; Nordic CML Study Group (NCMLSG). Impact of malignant stem cell burden on therapy outcome in newly diagnosed chronic myeloid leukemia patients. Leukemia. 2013 Jul;27(7):1520-6. doi: 10.1038/leu.2013.19. Epub 2013 Jan 18. PMID 23328954